CLINICAL TRIAL: NCT02643966
Title: Assessment of Periodic Screening of Women With Denser Breast Using WBUS and DBT (Also Known as "DBTUST-Dense Breast Tomosynthesis / Ultrasound Screening Trial")
Brief Title: Assessment of Periodic Screening of Women With Denser Breast Using WBUS and DBT
Acronym: DBTUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wendie Berg (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Wendie Berg, Professor of Radiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PRO14100275; R01CA187593-01A1 (NIH)
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: whole breast ultrasound; digital breast tomosynthesis; breast density; breast cancer screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole breast ultrasound (Experimental): All women will receive both 3D mammography and whole breast ultrasound for breast cancer screening; the order of interpretation will vary for each of two radiologists
  Interventions: Device: Whole breast ultrasound

INTERVENTIONS:
Device: Whole breast ultrasound — Breast cancer screening with whole breast ultrasound

SUMMARY:
The purpose of this study is to evaluate the role of technologist-performed whole breast ultrasound for detecting breast cancer in the screening population of women with dense breasts.

DETAILED DESCRIPTION:
This is a prospective study designed to evaluate the role of whole breast ultrasound (WBUS) in screening for breast cancer. In particular, there is interest in investigating the value of using WBUS as an adjunct (supplementary imaging) to Digital Breast Tomosynthesis (DBT) based screening of women with dense (heterogeneously or extremely dense) breasts or as a primary screening examination in this group of women. Women scheduled for their routine mammography that includes a DBT exam who agree to participate in the study and sign informed consent will undergo (at the same visit) DBT imaging as part of their clinical exam and whole breast ultrasound (WBUS) each year for three rounds of screening plus one year of follow-up. The DBT images and WBUS will be interpreted independently by two experienced radiologists under standard clinical screening procedures. One radiologist will interpret the DBT and the other radiologist will interpret the WBUS. Using a modified "LOGICAL OR" approach women/subjects may be recalled for further diagnostic work-up (examinations). If a subject is recalled, she will then follow the standard/routine clinical procedures for follow-up and the investigators will verify outcomes. If neither radiologist recalls the subject, then the subject will follow conventional management and the investigators will verify outcome. The findings from the DBT and WBUS examinations, as well as any resulting follow-up, will be collected, recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40 to 75 years of age with heterogeneously dense or extremely dense parenchyma by prior digital mammography report (i.e., "dense breasts"), presenting for routine annual mammography with digital breast tomosynthesis.

Exclusion Criteria:

* Known to be at high risk for breast cancer due to known or suspected pathologic BRCA mutation (i.e. first-degree relative with known mutation) or prior chest radiation therapy before age 30;
* No mammogram within the prior 3 years;
* Signs or symptoms of breast disease including lump, bloody or spontaneous clear nipple discharge, eczema of the nipple;
* Pregnancy or lactation within the prior 6 months;
* Plan to become pregnant in the next two years, as mammography is not typically performed for screening pregnant women;
* Breast implants, as assessment of breast density may be problematic;
* Recent prior breast surgery or breast biopsy or cyst aspiration within the prior 12 months;
* Prior or current malignancy other than the following: a) Breast cancer at least one year earlier (12 full months have elapsed since the last treatment surgery) with no known distant metastases and no known residual tumor; or b) Basal or squamous cell skin cancer or in situ cervical cancer or stage I thyroid cancer; or c) Other cancer for which the patient has been disease free for ≥ 5 years, with no recurrence of cancer in the last five years and no residual disease detected in the last five years.
* Screening contrast-enhanced MRI or 99mTc-sestamibi based imaging of the breast(s) within the prior 12 months or planned within the next two years, to avoid contamination of results;
* Unwilling or unable to provide consent.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6266 (Actual)
Dates: Start 2015-12; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendie Berg, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Weinstein Imaging Associates, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Berg WA, Zuley ML, Chang TS, Gizienski TA, Chough DM, Bohm-Velez M, Sharek DE, Straka MR, Hakim CM, Hartman JY, Harnist KS, Tyma CS, Kelly AE, Waheed U, Houshmand G, Nair BE, Shinde DD, Lu AH, Bandos AI, Berg JM, Lettiere NB, Ganott MA. Prospective Multicenter Diagnostic Performance of Technologist-Performed Screening Breast Ultrasound After Tomosynthesis in Women With Dense Breasts (the DBTUST). J Clin Oncol. 2023 May 1;41(13):2403-2415. doi: 10.1200/JCO.22.01445. Epub 2023 Jan 10. PMID 36626696

RESULTS

PARTICIPANT FLOW:
Period: First Screening Round
Arm/Group | Whole Breast Ultrasound
Started | 6266
Completed | 6178
Not Completed | 88
Not completed — ineligible | 1
Not completed — excluded from analysis | 2
Not completed — Lost to Follow-up | 56
Not completed — Withdrawal by Subject | 28
Not completed — Death | 1
Period: Between First and Second Screening
Arm/Group | Whole Breast Ultrasound
Started | 6178
Completed | 6020
Not Completed | 158
Not completed — Lost to Follow-up | 65
Not completed — Withdrawal by Subject | 82
Not completed — women who skipped year 2 exam | 11
Period: Second Screening Round
Arm/Group | Whole Breast Ultrasound
Started | 6020
Completed | 5937
Not Completed | 83
Not completed — Withdrawal by Subject | 20
Not completed — Lost to Follow-up | 57
Not completed — Physician Decision | 2
Not completed — Death | 4
Period: Between Second and Third Screening
Arm/Group | Whole Breast Ultrasound
Started | 5937
Completed | 5680
Not Completed | 257
Not completed — Lost to Follow-up | 75
Not completed — Death | 1
Not completed — Withdrawal by Subject | 181
Period: Third Screening Round
Arm/Group | Whole Breast Ultrasound
Started | 5680
Completed | 5437
Not Completed | 243
Not completed — PI excluded | 2
Not completed — Lost to Follow-up | 241

BASELINE CHARACTERISTICS:
Population: After exclusions, we analyzed the results from 6,179 women overall
Arm/Group | Whole Breast Ultrasound
Number analyzed (Participants) | 6179
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6179
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 6160
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 49
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 106
  White | 5991
  More than one race | 29
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6179
Breast Density [Count of Participants; unit: Participants]
  scattered | 203
  heterogeneously dense | 4989
  extremely dense | 987

OUTCOME MEASURES:

1. Primary Outcome: Cancer Yield Per 1,000
Description: Results from the first radiologist observer are presented
Time Frame: 3 Years
Population: Screens 2 & 3 include women who were analyzable after the end of Screening Round 2
Measure: Number (95% Confidence Interval); unit: Cancer yield per 1,000
Groups:
- Digital Breast Tomosynthesis (DBT): All women received both 3D mammography (DBT) and whole breast ultrasound (WBUS) for breast cancer screening. This Arm looks at the cancer yield per 1,000 for DBT alone.
- DBT and WBUS: All women received both 3D mammography (DBT) and whole breast ultrasound (WBUS) for breast cancer screening. This Arm looks at the cancer yield per 1,000 for DBT+WBUS.
Arm/Group | Digital Breast Tomosynthesis (DBT) | DBT and WBUS
Number analyzed (Participants) | 6178 | 6178
Cancer yield per 1,000
  Screen 1 | 5.0 [3.4 to 7.1] | 6.3 [4.5 to 8.6]
  Screens 2 & 3: number analyzed (Participants) | 5937 | 5937
  Screens 2 & 3 | 4.9 [4.0 to 5.9] | 5.9 [4.9 to 6.9]
Statistical Analysis 1: Comparison: Digital Breast Tomosynthesis (DBT) vs DBT and WBUS; The primary unit of analysis was the screening examination. A sample size of 16,700 screens (6,200 women, estimating 8%-10% loss to follow-up each year) was expected to provide 82% power to identify an added cancer detection rate (CDR) from US of 1.1/1,000. Screens were included for analysis if the patient was diagnosed with breast cancer or at least 10.5-month imaging or clinical follow-up (ie, at end of study participation) showed no evidence of breast cancer; Test type: Other — We compared DBT cancer yield per 1,000 for first observer (usual care) vs DBT and WBUS cancer yield per 1,000 for first observer for Year/Screen 1; p = 0.005, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; The 95% CIs for differences were estimated using nonparametric bootstrap approach on the basis of 10,000 replicates with women as resampling units; simple proportions = 1.3, 95% CI 2-sided [0.3 to 2.1]
Statistical Analysis 2: Comparison: Digital Breast Tomosynthesis (DBT) vs DBT and WBUS; [analysis description as in outcome 1, analysis 1]; Test type: Other — We compared DBT cancer yield per 1,000 for first observer (usual care) vs DBT and WBUS cancer yield per 1,000 for first observer for Years/Screens 2 & 3; p < 0.001, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; simple proportions = 1.0, 95% CI 2-sided [0.4 to 1.5]

2. Primary Outcome: Sensitivity (True Positive Rate)
Description: DBT true positive findings for first observer (usual care) vs DBT and WBUS true positive findings for first observer
Time Frame: 3 years
Population: Women diagnosed with cancer
Measure: Number (95% Confidence Interval); unit: percentage of participants with cancer
Groups:
- Digital Breast Tomosynthesis: All women received both 3D mammography and whole breast ultrasound for breast cancer screening; the order of interpretation varied for each of two radiologists. This Arm looks at the sensitivity of DBT alone for reader 1.
- DBT and WBUS: All women received both 3D mammography and whole breast ultrasound for breast cancer screening; the order of interpretation varied for each of two radiologists. This Arm looks at the sensitivity of DBT and WBUS for reader 1.
Arm/Group | Digital Breast Tomosynthesis | DBT and WBUS
Number analyzed (Participants) | 6178 | 6178
percentage of participants with cancer
  Year/Screen 1: number analyzed (Participants) | 45 | 45
  Year/Screen 1 | 68.9 [53.4 to 81.8] | 86.7 [73.2 to 95.0]
  Years/Screens 2 & 3: number analyzed (Participants) | 81 | 81
  Years/Screens 2 & 3 | 69.1 [57.9 to 78.9] | 82.7 [72.7 to 90.2]
Statistical Analysis 1: Comparison: Digital Breast Tomosynthesis vs DBT and WBUS; [analysis description as in outcome 1, analysis 1]; Test type: Other — We compared DBT true positive findings for first observer (usual care) vs DBT and WBUS true positive findings for first observer for Year/Screen 1; p = 0.005, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; simple proportions = 17.8, 95% CI 2-sided [4.4 to 31.1]
Statistical Analysis 2: Comparison: Digital Breast Tomosynthesis; The primary unit of analysis was the screening examination. A sample size of 16,700 screens (6,200 women, estimating 8%-10% loss to follow-up each year) was expected to provide 82% power to identify an added CDR from US of 1.1/1,000.Screens were included for analysis if the patient was diagnosed with breast cancer or at least 10.5-month imaging or clinical follow-up (ie, at end of study participation) showed no evidence of breast cancer; Test type: Other — We compared DBT true positive findings for first observer (usual care) vs DBT and WBUS true positive findings for first observer for Years/Screens 2 and 3; p < 0.001, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; simple proportions = 13.5, 95% CI 2-sided [4.9 to 22.3]

3. Secondary Outcome: Types of Abnormalities Detected by Ultrasound and Tomosynthesis
Description: Counts and percentages of participants diagnosed with cancer and detected by first observer with DBT only, DBT and WBUS, and WBUS only
Time Frame: 3 years
Population: Cancers detected by first observer for all 3 Screenings/Years combined
Measure: Count of Participants; unit: Participants
Groups:
- Digital Breast Tomosynthesis (DBT): All women received both 3D mammography (DBT) and whole breast ultrasound (WBUS) for breast cancer screening. This Arm looks at the number of cancers detected by first observer for DBT Alone.
- DBT and WBUS: All women received both 3D mammography (DBT) and whole breast ultrasound (WBUS) for breast cancer screening. This Arm looks at the number of cancers detected by first observer for DBT and WBUS.
- WBUS Only: All women received both 3D mammography (DBT) and whole breast ultrasound (WBUS) for breast cancer screening. This Arm looks at the number of cancers detected by first observer for WBUS alone.
Arm/Group | Digital Breast Tomosynthesis (DBT) | DBT and WBUS | WBUS Only
Number analyzed (Participants) | 17552 | 17552 | 17552
Participants
  No. of Cancers | 55 | 32 | 19
  No. of invasive cancers: number analyzed (Participants) | 55 | 32 | 19
  No. of invasive cancers | 32 | 31 | 16
  No. of Node-positive among available staging: number analyzed (Participants) | 29 | 29 | 16
  No. of Node-positive among available staging | 3 | 5 | 3

4. Primary Outcome: False-positive Recall Rate
Description: DBT false-positive findings for first observer (usual care) vs DBT and WBUS false positive findings for first observer
Time Frame: 3 years
Population: Women who did not have a cancer diagnosis
Measure: Number (95% Confidence Interval); unit: percent of participants without cancer
Groups:
- Digital Breast Tomosynthesis: All women received both 3D mammography and whole breast ultrasound for breast cancer screening; the order of interpretation varied for each of two radiologists. This Arm looks at the false-positive recall rate of DBT alone for reader 1.
- DBT and WBUS: All women received both 3D mammography and whole breast ultrasound for breast cancer screening; the order of interpretation varied for each of two radiologists. This arm looks at the false-positive recall rate of DBT and WBUS for reader 1.
Arm/Group | Digital Breast Tomosynthesis | DBT and WBUS
Number analyzed (Participants) | 6178 | 6178
percent of participants without cancer
  Year/Screen 1: number analyzed (Participants) | 6133 | 6133
  Year/Screen 1 | 7.0 [6.4 to 7.7] | 11.5 [10.7 to 12.3]
  Years/Screens 2 & 3: number analyzed (Participants) | 5856 | 5856
  Years/Screens 2 & 3 | 5.9 [5.5 to 6.4] | 9.7 [9.1 to 10.2]
Statistical Analysis 1: Comparison: Digital Breast Tomosynthesis vs DBT and WBUS; Test type: Other — We compared DBT false positive findings for first observer (usual care) vs DBT and WBUS false positive findings for first observer for Year/Screen 1; p < 0.001, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Slope = 4.5, 95% CI 2-sided [3.8 to 5.1]
Statistical Analysis 2: Comparison: Digital Breast Tomosynthesis vs DBT and WBUS; Test type: Other — We compared DBT false positive findings for first observer (usual care) vs DBT and WBUS false positive findings for first observer for Years/Screens 2 & 3; p < 0.001, nonparametric bootstrap approach — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; simple proportions = 3.7, 95% CI 2-sided [3.3 to 4.1]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Whole Breast Ultrasound
All-Cause Mortality (participants affected / at risk) | 6/6266
Serious Adverse Events (participants affected / at risk) | 0/6266
Other Adverse Events (participants affected / at risk) | 0/6266

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02643966/Prot_SAP_000.pdf